CLINICAL TRIAL: NCT01803282
Title: A Phase 1 Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of GS-5745 as Monotherapy and in Combination With Chemotherapy in Subjects With Advanced Solid Tumors
Brief Title: Study to Evaluate the Safety and Tolerability of Andecaliximab as Monotherapy and in Combination With Chemotherapy in Participants With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: GS-US-296-0101
Record Dates: First submitted 2013-02-27; First posted 2013-03-04 (Estimated); Results first posted 2020-05-04 (Actual); Last update posted 2020-06-02 (Actual); Status verified 2020-05

CONDITIONS: Pancreatic Cancer; Non-small Cell Lung Cancer; Esophagogastric Cancer; Colorectal Cancer; Breast Cancer
Keywords: Solid Tumor
MeSH Terms: conditions — Pancreatic Neoplasms; Carcinoma, Non-Small-Cell Lung; Colorectal Neoplasms; Breast Neoplasms | interventions — andecaliximab; Gemcitabine; 130-nm albumin-bound paclitaxel; Carboplatin; Pemetrexed; Leucovorin; Oxaliplatin; Fluorouracil; Bevacizumab; Irinotecan; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (12):
- Part A: ADX 200 mg (Experimental): Participants with advanced solid tumors who fail or are intolerant to standard therapy or for whom no standard therapy exists, will receive 200 mg ADX as monotherapy via IV infusion (approximately 30 minutes) every 2 weeks until disease progression, unacceptable toxicity, withdrawal of consent, or other reasons prespecified in the protocol for discontinuation of study drug.
  Interventions: Drug: Andecaliximab
- Part A: ADX 600 mg (Experimental): Participants with advanced solid tumors who fail or are intolerant to standard therapy or for whom no standard therapy exists, will receive 600 mg ADX as monotherapy via IV infusion (approximately 30 minutes) every 2 weeks until disease progression, unacceptable toxicity, withdrawal of consent, or other reasons prespecified in the protocol for discontinuation of study drug.
  Interventions: Drug: Andecaliximab
- Part A: ADX 1800 mg (Experimental): Participants with advanced solid tumors who fail or are intolerant to standard therapy or for whom no standard therapy exists, will receive 1800 mg ADX as monotherapy via IV infusion (approximately 30 minutes) every 2 weeks until disease progression, unacceptable toxicity, withdrawal of consent, or other reasons prespecified in the protocol for discontinuation of study drug
  Interventions: Drug: Andecaliximab
- Part B: PAC, ADX 800 mg (Experimental): Participants with PAC will receive ADX 800 mg every 2 weeks via IV infusion in addition to the 28-day cycle chemotherapy (gemcitabine and nab paclitaxel, on Days 1, 8, and 15) until disease progression, unacceptable toxicity, withdrawal of consent, or other reasons prespecified in the protocol for discontinuation of study drug.
  Interventions: Drug: Andecaliximab; Drug: Gemcitabine; Drug: Nab-paclitaxel
- Part B: LAC, ADX 1200 mg (Experimental): Participants with lung adenocarcinoma (LAC) will receive ADX 1200 mg every 3 weeks via IV infusion in addition to the 21-day cycle chemotherapy (carboplatin and pemetrexed, on Day 1) until disease progression, unacceptable toxicity, withdrawal of consent, or other reasons prespecified in the protocol for discontinuation of study drug.
  Interventions: Drug: Andecaliximab; Drug: Carboplatin; Drug: Pemetrexed
- Part B: LSC, ADX 1200 mg (Experimental): Participants with lung squamous cell carcinoma (LSC) will receive ADX 1200 mg every 3 weeks via IV infusion in addition to the 21-day cycle chemotherapy (carboplatin and paclitaxel, on Day 1) until disease progression, unacceptable toxicity, withdrawal of consent, or other reasons prespecified in the protocol for discontinuation of study drug.
  Interventions: Drug: Andecaliximab; Drug: Carboplatin; Drug: Paclitaxel
- Part B: EGC, ADX 800 mg (Experimental): Participants with esophagogastric adenocarcinoma (EGC) will receive ADX 800 mg every 2 weeks via IV infusion in addition to the 28-day cycle chemotherapy (leucovorin+oxaliplatin+5-fluorouracil {5-FU} [mFOLFOX6], on Days 1 and 15) until disease progression, unacceptable toxicity, withdrawal of consent, or other reasons prespecified in the protocol for discontinuation of study drug.
  Interventions: Drug: Andecaliximab; Drug: Leucovorin; Drug: Oxaliplatin; Drug: 5-FU
- Part B: FL CRC, ADX 800 mg+BEV 5 mg/kg (Experimental): Participants with colorectal cancer (CRC) will receive first-line (FL) treatment with ADX 800 mg every 2 weeks via IV infusion in addition to the 28-day cycle chemotherapy (mFOLFOX6 and bevacizumab 5 mg/kg, on Days 1 and 15) until disease progression, unacceptable toxicity, withdrawal of consent, or other reasons prespecified in the protocol for discontinuation of study drug.
  Interventions: Drug: Andecaliximab; Drug: Leucovorin; Drug: Oxaliplatin; Drug: 5-FU; Drug: Bevacizumab
- Part B: FL CRC, ADX 800 mg+BEV 10 mg/kg (Experimental): Participants with CRC will receive FL treatment with ADX 800 mg every 2 weeks via IV infusion in addition to the 28-day cycle chemotherapy (mFOLFOX6 and bevacizumab 10 mg/kg, on Days 1 and 15) until disease progression, unacceptable toxicity, withdrawal of consent, or other reasons prespecified in the protocol for discontinuation of study drug.
  Interventions: Drug: Andecaliximab; Drug: Leucovorin; Drug: Oxaliplatin; Drug: 5-FU; Drug: Bevacizumab
- Part B: SL CRC, ADX 800 mg+BEV 5 mg/kg (Experimental): Participants with CRC will receive second-line (SL) treatment with ADX 800 mg every 2 weeks via IV infusion in addition to the 28-day cycle chemotherapy (leucovorin+irinotecan+5-FU [FOLFIRI] and bevacizumab 5 mg/kg, on Days 1 and 15) until disease progression, unacceptable toxicity, withdrawal of consent, or other reasons prespecified in the protocol for discontinuation of study drug.
  Interventions: Drug: Andecaliximab; Drug: Leucovorin; Drug: 5-FU; Drug: Bevacizumab; Drug: Irinotecan
- Part B: SL CRC, ADX 800 mg+BEV 10 mg/kg (Experimental): Participants with CRC will receive SL treatment with ADX 800 mg every 2 weeks via IV infusion in addition to the 28-day cycle chemotherapy (FOLFIRI and bevacizumab 10 mg/kg, on Days 1 and 15) until disease progression, unacceptable toxicity, withdrawal of consent, or other reasons prespecified in the protocol for discontinuation of study drug.
  Interventions: Drug: Andecaliximab; Drug: Leucovorin; Drug: 5-FU; Drug: Bevacizumab; Drug: Irinotecan
- Part B: BRCA, ADX 800 mg (Experimental): Participants with breast cancer (BRCA) will receive ADX 800 mg every 2 weeks via IV infusion in addition to the 28-day cycle chemotherapy (paclitaxel, on Days 1, 8, and 15) until disease progression, unacceptable toxicity, withdrawal of consent, or other reasons prespecified in the protocol for discontinuation of study drug.
  Interventions: Drug: Andecaliximab; Drug: Paclitaxel

INTERVENTIONS:
Drug: Andecaliximab — Administered intravenous infusion
  Other Names: GS-5745
Drug: Gemcitabine — Administered intravenously on Days 1, 8, and 15 of each 28-day treatment cycle
  Arms: Part B: PAC, ADX 800 mg
Drug: Nab-paclitaxel — Administered intravenously on Days 1, 8, and 15 of each 28-day treatment cycle
  Arms: Part B: PAC, ADX 800 mg
Drug: Carboplatin — Administered intravenously on Day 1 of each 21-day treatment cycle
  Arms: Part B: LAC, ADX 1200 mg; Part B: LSC, ADX 1200 mg
Drug: Pemetrexed — Administered intravenously on Day 1 of each 21-day treatment cycle
  Arms: Part B: LAC, ADX 1200 mg
Drug: Leucovorin — Administered intravenously on Days 1 and 15 of each 28-day treatment cycle
  Arms: Part B: EGC, ADX 800 mg; Part B: FL CRC, ADX 800 mg+BEV 10 mg/kg; Part B: FL CRC, ADX 800 mg+BEV 5 mg/kg; Part B: SL CRC, ADX 800 mg+BEV 10 mg/kg; Part B: SL CRC, ADX 800 mg+BEV 5 mg/kg
Drug: Oxaliplatin — Administered intravenously on Days 1 and 15 of each 28-day treatment cycle
  Arms: Part B: EGC, ADX 800 mg; Part B: FL CRC, ADX 800 mg+BEV 10 mg/kg; Part B: FL CRC, ADX 800 mg+BEV 5 mg/kg
Drug: 5-FU — Administered intravenously on Days 1 and 15 of each 28-day treatment cycle
  Arms: Part B: EGC, ADX 800 mg; Part B: FL CRC, ADX 800 mg+BEV 10 mg/kg; Part B: FL CRC, ADX 800 mg+BEV 5 mg/kg; Part B: SL CRC, ADX 800 mg+BEV 10 mg/kg; Part B: SL CRC, ADX 800 mg+BEV 5 mg/kg
Drug: Bevacizumab — Administered intravenously on Days 1 and 15 of each 28-day treatment cycle
  Arms: Part B: FL CRC, ADX 800 mg+BEV 10 mg/kg; Part B: FL CRC, ADX 800 mg+BEV 5 mg/kg; Part B: SL CRC, ADX 800 mg+BEV 10 mg/kg; Part B: SL CRC, ADX 800 mg+BEV 5 mg/kg
Drug: Irinotecan — Administered intravenously on Days 1 and 15 of each 28-day treatment cycle
  Arms: Part B: SL CRC, ADX 800 mg+BEV 10 mg/kg; Part B: SL CRC, ADX 800 mg+BEV 5 mg/kg
Drug: Paclitaxel — Administered intravenously on Days 1, 8 and 15 of each 28-day treatment cycle (Breast cancer) or on Day 1 of each 21-day treatment cycle (NSCLC)
  Arms: Part B: BRCA, ADX 800 mg; Part B: LSC, ADX 1200 mg

SUMMARY:
The primary objective of the study is to determine the maximum tolerated dose of andecaliximab monotherapy and to evaluate the safety and tolerability of andecaliximab (formerly GS-5745) alone and in combination with chemotherapy.

The study consists of 2 parts (Parts A and B). Participants can only qualify for and participate in 1 part.

Part A is a sequential dose escalation to determine the maximum tolerated dose of andecaliximab in participants with advanced solid tumors that are refractory to or intolerant to standard therapy or for which no standard therapy exists. In Part A, participants will receive andecaliximab only.

Part B is a dose expansion to obtain additional safety and tolerability data for andecaliximab in participants with advanced pancreatic adenocarcinoma, lung adenocarcinoma, lung squamous cell carcinoma, esophagogastric adenocarcinoma, colorectal cancer, or breast cancer. In Part B, participants will receive andecaliximab in combination with standard-of-care chemotherapy.

ELIGIBILITY:
Key Inclusion Criteria:

* Part A: histologically or cytologically confirmed advanced malignant solid tumor that is refractory to or intolerant of standard therapy or for which no standard therapy is available
* Part B: Pancreatic Adenocarcinoma

  * Presence of histologically confirmed inoperable locally advanced or metastatic pancreatic adenocarcinoma
* Part B: NSCLC

  * Stage IIIB with malignant pleural effusion/pleural seeding or stage IV histologically confirmed NSCLC
  * Absence of known epidermal growth factor receptor (EGFR) mutation
  * Absence of known translocation or inversion events involving the ALK gene locus (resulting in EML4-ALK fusion)
* Part B: Esophagogastric Adenocarcinoma:

  * Histologically confirmed inoperable advanced gastric adenocarcinoma (including adenocarcinoma of the gastrooesophageal junction) or relapsed gastric adenocarcinoma
  * Human epidermal growth factor receptor 2 (HER2)-negative tumor (primary tumor or metastatic lesion)
* Part B: First-Line Colorectal Cancer

  * Histologically confirmed inoperable advanced adenocarcinoma of the colon or rectum
  * Radiographically measureable disease
  * No prior cytotoxic chemotherapy to treat their metastatic disease
* Part B: Second-Line Colorectal Cancer

  * Histologically confirmed inoperable advanced adenocarcinoma of the colon or rectum
  * Radiographically measureable disease
  * Received first-line combination therapy containing oxaliplatin and fluoropyrimidine with or without bevacizumab for metastatic disease with documented evidence of disease progression during or after treatment completion
* Part B: Breast Cancer

  * Histologically or cytologically confirmed metastatic breast cancer
  * Radiographically measureable disease
  * Previous hormonal therapy for metastatic breast cancer or cytotoxic adjuvant chemotherapy is allowed
  * Treatment with weekly single-agent paclitaxel is appropriate in the opinion of the treating physician
  * HER-2 negative tumor (primary tumor or metastatic lesion)
* Adequate organ function

Key Exclusion Criteria:

* Pregnant or lactating
* Individuals with known central nervous system (CNS) metastases, unless metastases are treated and stable and the individual does not require systemic steroids
* Myocardial infarction, symptomatic congestive heart failure, unstable angina, or serious uncontrolled cardiac arrhythmia within the last 6 months
* Anti-tumor therapy within 28 days of study drug dosing; concurrent use of hormone therapy for breast or prostate cancer is permitted

Note: Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 236 (Actual)
Dates: Start 2013-03-29 (Actual); Primary Completion 2019-04-23 (Actual); Study Completion 2019-04-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gilead Study Director, Study Director — Gilead Sciences
Locations (18):
- United States (18):
  - Alabama Oncology, Birmingham, Alabama
  - Pinnacle Oncology Hematology, Scottsdale, Arizona
  - Comprehensive Blood and Cancer Center, Bakersfield, California
  - San Diego Pacific Oncology and Hematology Associates, Inc., Encinitas, California
  - University of Southern California (USC), Los Angeles, California
  - California Pacific Medical Center, San Francisco, California
  - UCLA Medical Center, Santa Monica, California
  - Florida Cancer Specialists, Sarasota, Florida
  - Parkview Research Center, Fort Wayne, Indiana
  - Indiana University Health Goshen Center for Cancer Care, Goshen, Indiana
  - Washington University School of Medicine, St Louis, Missouri
  - Cornell University, New York, New York
  - Greenville Health System, Institute for Translational Oncology Research, Greenville, South Carolina
  - Sarah Cannon Research Institute, Nashville, Tennessee
  - Vanderbilt, Nashville, Tennessee
  - UT Southwestern, Dallas, Texas
  - University of Utah, Salt Lake City, Utah
  - Northwest Medical Specialties, Tacoma, Washington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Shah MA, Starodub A, Sharma S, Berlin J, Patel M, Wainberg ZA, Chaves J, Gordon M, Windsor K, Brachmann CB, Huang X, Vosganian G, Maltzman JD, Smith V, Silverman JA, Lenz HJ, Bendell JC. Andecaliximab/GS-5745 Alone and Combined with mFOLFOX6 in Advanced Gastric and Gastroesophageal Junction Adenocarcinoma: Results from a Phase I Study. Clin Cancer Res. 2018 Aug 15;24(16):3829-3837. doi: 10.1158/1078-0432.CCR-17-2469. Epub 2018 Apr 24. PMID 29691300
- [Result] Lenz H, Park H, Shah MA, Berlin JD, Bruetman D, Chaves J, et al. Results of a phase I study of andecaliximab in combination with mFOLFOX6 and bevacizumab in patients with previously untreated metastatic colorectal cancer. Annals of Oncology (2018) 29 (suppl_8): viii150-viii204
- [Result] Wainberg Z, Bendell J, Lenz H, Baron A, Berlin J, Bessudo A, et al. Results from a phase I study of andecaliximab in combination with FOLFIRI and bevacizumab in patients with second line metastatic colorectal cancer. Journal of Clinical Oncology 36, no. 15_suppl (May 20, 2018) 3578-3578
- [Result] Bendell J, Patel M, Brachmann C, Huang X, Maltzman J, Smith V, et al. Updated results of a phase 1 study combining the matrix metalloproteinase 9 inhibitor GS-5745 with gemcitabine and nab-paclitaxel in patients with advanced pancreatic cancer [Abstract 363] 2017 American Society of Clinical Oncology Gastrointestinal Cancers Symposium
- [Result] Brachmann C, Zhang Y, Zavodovskaya M, Hu J, Maltzman J, Smith V, et al. Evaluating collagen neoepitopes as pharmacodynamic biomarkers of GS-5745, an MMP9 inhibitor, in advanced gastric cancer [Abstract 58] 2017 American Society of Clinical Oncology Gastrointestinal Cancers Symposium
- [Result] Juric V, Mikels-Vigdal A, O'Sullivan C, Greenstein A, Stefanutti E, Barry-Hamilton V, et al. Inhibition of MMP9 improves anti-tumor immunity by changing the tumor microenvironment to promote T cell trafficking and activation. [Abstract 653/27]. 2017 American Association for Cancer Research Annual Meeting 110th Annual Meeting; 2017 01 April-05 April; Washington, DC
- [Result] Zavodovskaya M, Zhang Y, Xiao Y, Maltzman J, Smith V, Brachmann C, et al. Exploratory Serum Biomarker Analysis in Gastric Cancer Patients Treated with GS-5745, an MMP9 Inhibitor, in Combination with mFOLFOX6 [Abstract 4463/24]. 2017 American Association for Cancer Research Annual Meeting 110th Annual Meeting; 2017 01 April-05 April; Washington, DC
- [Result] Bendell J, Huang X, Smith V, Maltzman J, Starodub A. Results of a phase I study of GS-5745 in combination with gemcitabine and nab-paclitaxel in patients (pts) with advanced pancreatic cancer [abstract e15683] 2016. J Clin Oncol 34 supplemental
- [Result] Shah M, Starodub A, Wainberg Z, Smith V, Maltzman J, Bendell J. Results of a phase I study of GS-5745 in combination with mFOLFOX in patients with advanced unresectable gastric / GE junction tumors [Poster 4033]. American Society of Clinical Oncology (ASCO) 52nd Annual Meeting; 2016 03 June- 07 June; Chicago, IL
- [Result] Bendell J, Starodub A, Sharma S, Wainberg Z, Shah M, Thai D. Phase I Study of GS-5745 Alone and in Combination with Chemotherapy in Patients with Advanced Solid Tumors [Poster 4030]. American Society of Clinical Oncology (ASCO) 51st Annual Meeting; 2015 29 May-02 June; Chicago, IL
- [Result] Marshall DC, Lyman SK, McCauley S, Kovalenko M, Spangler R, Liu C, Lee M, O'Sullivan C, Barry-Hamilton V, Ghermazien H, Mikels-Vigdal A, Garcia CA, Jorgensen B, Velayo AC, Wang R, Adamkewicz JI, Smith V. Selective Allosteric Inhibition of MMP9 Is Efficacious in Preclinical Models of Ulcerative Colitis and Colorectal Cancer. PLoS One. 2015 May 11;10(5):e0127063. doi: 10.1371/journal.pone.0127063. eCollection 2015. PMID 25961845

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at study sites in the United States. The first participant was screened on 29 March 2013. The last study visit occurred on 23 April 2019.
Pre-assignment Details: 280 participants were screened.
Groups:
- Part A: ADX 200 mg: Participants with advanced solid tumors who had failed or were intolerant to standard therapy or for whom no standard therapy existed, received 200 mg andecaliximab (ADX) as monotherapy via intravenous (IV) infusion (approximately 30 minutes) every 2 weeks until disease progression, unacceptable toxicity, withdrawal of consent, or other reasons prespecified in the protocol for discontinuation of study drug.
- Part A: ADX 600 mg: Participants with advanced solid tumors who had failed or were intolerant to standard therapy or for whom no standard therapy existed, received 600 mg ADX as monotherapy via IV infusion (approximately 30 minutes) every 2 weeks until disease progression, unacceptable toxicity, withdrawal of consent, or other reasons prespecified in the protocol for discontinuation of study drug.
- Part A: ADX 1800 mg: Participants with advanced solid tumors who had failed or were intolerant to standard therapy or for whom no standard therapy existed, received 1800 mg ADX as monotherapy via IV infusion (approximately 30 minutes) every 2 weeks until disease progression, unacceptable toxicity, withdrawal of consent, or other reasons prespecified in the protocol for discontinuation of study drug.
- Part B: PAC, ADX 800 mg: Participants with pancreatic adenocarcinoma (PAC) received ADX 800 mg every 2 weeks via IV infusion in addition to the 28-day cycle chemotherapy (gemcitabine and nab paclitaxel, on Days 1, 8, and 15) until disease progression, unacceptable toxicity, withdrawal of consent, or other reasons prespecified in the protocol for discontinuation of study drug.
- Part B: LAC, ADX 1200 mg: Participants with lung adenocarcinoma (LAC) received ADX 1200 mg every 3 weeks via IV infusion in addition to the 21-day cycle chemotherapy (carboplatin and pemetrexed, on Day 1) until disease progression, unacceptable toxicity, withdrawal of consent, or other reasons prespecified in the protocol for discontinuation of study drug.
- Part B: LSC, ADX 1200 mg: Participants with lung squamous cell carcinoma (LSC) received ADX 1200 mg every 3 weeks via IV infusion in addition to the 21-day cycle chemotherapy (carboplatin and paclitaxel, on Day 1) until disease progression, unacceptable toxicity, withdrawal of consent, or other reasons prespecified in the protocol for discontinuation of study drug.
- Part B: EGC, ADX 800 mg: Participants with esophagogastric adenocarcinoma (EGC) received ADX 800 mg every 2 weeks via IV infusion in addition to the 28-day cycle chemotherapy (leucovorin+oxaliplatin+5-fluorouracil {5-FU} [mFOLFOX6], on Days 1 and 15) until disease progression, unacceptable toxicity, withdrawal of consent, or other reasons prespecified in the protocol for discontinuation of study drug.
- Part B: FL CRC, ADX 800 mg+BEV 5 mg/kg: Participants with colorectal cancer (CRC) received first-line (FL) treatment with ADX 800 mg every 2 weeks via IV infusion in addition to the 28-day cycle chemotherapy (mFOLFOX6 and bevacizumab 5 mg/kg, on Days 1 and 15) until disease progression, unacceptable toxicity, withdrawal of consent, or other reasons prespecified in the protocol for discontinuation of study drug.
- Part B: FL CRC, ADX 800 mg+BEV 10 mg/kg: Participants with CRC received FL treatment with ADX 800 mg every 2 weeks via IV infusion in addition to the 28-day cycle chemotherapy (mFOLFOX6 and bevacizumab 10 mg/kg, on Days 1 and 15) until disease progression, unacceptable toxicity, withdrawal of consent, or other reasons prespecified in the protocol for discontinuation of study drug.
- Part B: SL CRC, ADX 800 mg+BEV 5 mg/kg: Participants with CRC received second-line (SL) treatment with ADX 800 mg every 2 weeks via IV infusion in addition to the 28-day cycle chemotherapy (leucovorin+irinotecan+5-FU [FOLFIRI] and bevacizumab 5 mg/kg, on Days 1 and 15) until disease progression, unacceptable toxicity, withdrawal of consent, or other reasons prespecified in the protocol for discontinuation of study drug.
- Part B: SL CRC, ADX 800 mg+BEV 10 mg/kg: Participants with CRC received SL treatment with ADX 800 mg every 2 weeks via IV infusion in addition to the 28-day cycle chemotherapy (FOLFIRI and bevacizumab 10 mg/kg, on Days 1 and 15) until disease progression, unacceptable toxicity, withdrawal of consent, or other reasons prespecified in the protocol for discontinuation of study drug.
- Part B: BRCA, ADX 800 mg: Participants with breast cancer (BRCA) received ADX 800 mg every 2 weeks via IV infusion in addition to the 28-day cycle chemotherapy (paclitaxel, on Days 1, 8, and 15) until disease progression, unacceptable toxicity, withdrawal of consent, or other reasons prespecified in the protocol for discontinuation of study drug.
Period: Overall Study
Arm/Group | Part A: ADX 200 mg | Part A: ADX 600 mg | Part A: ADX 1800 mg | Part B: PAC, ADX 800 mg | Part B: LAC, ADX 1200 mg | Part B: LSC, ADX 1200 mg | Part B: EGC, ADX 800 mg | Part B: FL CRC, ADX 800 mg+BEV 5 mg/kg | Part B: FL CRC, ADX 800 mg+BEV 10 mg/kg | Part B: SL CRC, ADX 800 mg+BEV 5 mg/kg | Part B: SL CRC, ADX 800 mg+BEV 10 mg/kg | Part B: BRCA, ADX 800 mg
Started | 4 | 3 | 6 | 36 | 11 | 10 | 41 | 46 | 11 | 45 | 8 | 15
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 4 | 3 | 6 | 36 | 11 | 10 | 41 | 46 | 11 | 45 | 8 | 15
Not completed — Progressive Disease | 4 | 3 | 6 | 22 | 5 | 8 | 23 | 24 | 3 | 29 | 6 | 11
Not completed — Death | 0 | 0 | 0 | 0 | 2 | 1 | 1 | 5 | 1 | 1 | 0 | 0
Not completed — Withdrew Consent | 0 | 0 | 0 | 6 | 1 | 0 | 8 | 3 | 1 | 5 | 0 | 1
Not completed — Investigator's Discretion | 0 | 0 | 0 | 7 | 2 | 1 | 7 | 10 | 6 | 7 | 1 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 1 | 0 | 3
Not completed — Non-Compliance with Study Drug | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Unknown Reason | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Specified Criteria for Withdrawal | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Not completed — Enrolled but Never Treated | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The Safety Analysis Set included all participants who received at least 1 infusion at any dose level of study drug (ADX).
Groups:
- Part A: ADX 200 mg: Participants with advanced solid tumors who had failed or were intolerant to standard therapy or for whom no standard therapy existed, received 200 mg ADX as monotherapy via IV infusion (approximately 30 minutes) every 2 weeks until disease progression, unacceptable toxicity, withdrawal of consent, or other reasons prespecified in the protocol for discontinuation of study drug.
- Part B: PAC, ADX 800 mg: Participants with PAC received ADX 800 mg every 2 weeks via IV infusion in addition to the 28-day cycle chemotherapy (gemcitabine and nab paclitaxel, on Days 1, 8, and 15) until disease progression, unacceptable toxicity, withdrawal of consent, or other reasons prespecified in the protocol for discontinuation of study drug.
- Part B: LAC, ADX 1200 mg: Participants with LAC received ADX 1200 mg every 3 weeks via IV infusion in addition to the 21-day cycle chemotherapy (carboplatin and pemetrexed, on Day 1) until disease progression, unacceptable toxicity, withdrawal of consent, or other reasons prespecified in the protocol for discontinuation of study drug.
- Part B: LSC, ADX 1200 mg: Participants with LSC received ADX 1200 mg every 3 weeks via IV infusion in addition to the 21-day cycle chemotherapy (carboplatin and paclitaxel, on Day 1) until disease progression, unacceptable toxicity, withdrawal of consent, or other reasons prespecified in the protocol for discontinuation of study drug.
- Part B: EGC, ADX 800 mg: Participants with EGC received ADX 800 mg every 2 weeks via IV infusion in addition to the 28-day cycle chemotherapy (mFOLFOX6, on Days 1 and 15) until disease progression, unacceptable toxicity, withdrawal of consent, or other reasons prespecified in the protocol for discontinuation of study drug.
- Part B: FL CRC, ADX 800 mg+BEV 5 mg/kg: Participants with CRC received FL treatment with ADX 800 mg every 2 weeks via IV infusion in addition to the 28-day cycle chemotherapy (mFOLFOX6 and bevacizumab 5 mg/kg, on Days 1 and 15) until disease progression, unacceptable toxicity, withdrawal of consent, or other reasons prespecified in the protocol for discontinuation of study drug.
- Part B: SL CRC, ADX 800 mg+BEV 5 mg/kg: Participants with CRC received SL treatment with ADX 800 mg every 2 weeks via IV infusion in addition to the 28-day cycle chemotherapy (FOLFIRI and bevacizumab 5 mg/kg, on Days 1 and 15) until disease progression, unacceptable toxicity, withdrawal of consent, or other reasons prespecified in the protocol for discontinuation of study drug.
- Part B: BRCA, ADX 800 mg: Participants with BRCA received ADX 800 mg every 2 weeks via IV infusion in addition to the 28-day cycle chemotherapy (paclitaxel, on Days 1, 8, and 15) until disease progression, unacceptable toxicity, withdrawal of consent, or other reasons prespecified in the protocol for discontinuation of study drug.
- Total: Total of all reporting groups
Arm/Group | Part A: ADX 200 mg | Part A: ADX 600 mg | Part A: ADX 1800 mg | Part B: PAC, ADX 800 mg | Part B: LAC, ADX 1200 mg | Part B: LSC, ADX 1200 mg | Part B: EGC, ADX 800 mg | Part B: FL CRC, ADX 800 mg+BEV 5 mg/kg | Part B: FL CRC, ADX 800 mg+BEV 10 mg/kg | Part B: SL CRC, ADX 800 mg+BEV 5 mg/kg | Part B: SL CRC, ADX 800 mg+BEV 10 mg/kg | Part B: BRCA, ADX 800 mg | Total
Number analyzed (Participants) | 4 | 3 | 6 | 36 | 10 | 10 | 40 | 45 | 11 | 44 | 8 | 15 | 232
Age, Customized [Count of Participants; unit: Participants]
  Age: < 65 years | 2 | 0 | 4 | 15 | 2 | 4 | 25 | 26 | 8 | 33 | 4 | 10 | 133
  Age: ≥ 65 years | 2 | 3 | 2 | 21 | 8 | 6 | 15 | 19 | 3 | 11 | 4 | 5 | 99
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 2 | 10 | 7 | 4 | 9 | 19 | 3 | 25 | 2 | 13 | 95
  Male | 3 | 3 | 4 | 26 | 3 | 6 | 31 | 26 | 8 | 19 | 6 | 2 | 137
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Ethnicity: Hispanic or Latino | 0 | 0 | 0 | 4 | 0 | 1 | 4 | 4 | 0 | 4 | 0 | 2 | 19
  Ethnicity: Not Hispanic or Latino | 4 | 3 | 6 | 32 | 10 | 9 | 30 | 39 | 10 | 39 | 8 | 12 | 202
  Ethnicity: Not Permitted | 0 | 0 | 0 | 0 | 0 | 0 | 6 | 2 | 1 | 1 | 0 | 1 | 11
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: American Indian or Alaska Native | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 3
  Race: Asian | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 2 | 0 | 0 | 4
  Race: Black or African American | 0 | 0 | 1 | 0 | 1 | 3 | 1 | 6 | 2 | 2 | 1 | 1 | 18
  Race: Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Race: White | 3 | 3 | 5 | 33 | 9 | 5 | 31 | 35 | 8 | 35 | 6 | 12 | 185
  Race: Not Permitted | 1 | 0 | 0 | 0 | 0 | 0 | 6 | 3 | 0 | 2 | 0 | 1 | 13
  Race: Other | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 1 | 1 | 2 | 1 | 1 | 9

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Experiencing Treatment-Emergent Adverse Events
Time Frame: Part A: First dose date up to 32 weeks plus 30 days; Part B: First dose date up to 181 weeks plus 30 days
Population: as for baseline characteristics
Measure: Number; unit: percentage of participants
Arm/Group | Part A: ADX 200 mg | Part A: ADX 600 mg | Part A: ADX 1800 mg | Part B: PAC, ADX 800 mg | Part B: LAC, ADX 1200 mg | Part B: LSC, ADX 1200 mg | Part B: EGC, ADX 800 mg | Part B: FL CRC, ADX 800 mg+BEV 5 mg/kg | Part B: FL CRC, ADX 800 mg+BEV 10 mg/kg | Part B: SL CRC, ADX 800 mg+BEV 5 mg/kg | Part B: SL CRC, ADX 800 mg+BEV 10 mg/kg | Part B: BRCA, ADX 800 mg
Number analyzed (Participants) | 4 | 3 | 6 | 36 | 10 | 10 | 40 | 45 | 11 | 44 | 8 | 15
percentage of participants | 100.0 | 100.0 | 83.3 | 100.0 | 100.0 | 100.0 | 100.0 | 100.0 | 100.0 | 100.0 | 100.0 | 100.0

2. Primary Outcome: Percentage of Participants Experiencing Laboratory Abnormalities
Description: Treatment-emergent laboratory abnormalities were defined as values that increase at least one toxicity grade from baseline. Participants with any laboratory abnormality were reported.
Time Frame: Part A: First dose date up to 32 weeks plus 30 days; Part B: First dose date up to 181 weeks plus 30 days
Population: Participants in the Safety Analysis Set were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | Part A: ADX 200 mg | Part A: ADX 600 mg | Part A: ADX 1800 mg | Part B: PAC, ADX 800 mg | Part B: LAC, ADX 1200 mg | Part B: LSC, ADX 1200 mg | Part B: EGC, ADX 800 mg | Part B: FL CRC, ADX 800 mg+BEV 5 mg/kg | Part B: FL CRC, ADX 800 mg+BEV 10 mg/kg | Part B: SL CRC, ADX 800 mg+BEV 5 mg/kg | Part B: SL CRC, ADX 800 mg+BEV 10 mg/kg | Part B: BRCA, ADX 800 mg
Number analyzed (Participants) | 4 | 3 | 6 | 36 | 10 | 10 | 40 | 45 | 11 | 44 | 8 | 15
percentage of participants
  Any Laboratory abnormalities: Hematology | 0.0 | 33.3 | 33.3 | 97.2 | 90.0 | 80.0 | 87.5 | 84.4 | 90.9 | 95.5 | 100.0 | 86.7
  Any Laboratory abnormalities: Serum Chemistry | 100.0 | 66.7 | 83.3 | 88.9 | 60.0 | 70.0 | 87.5 | 95.6 | 81.8 | 86.4 | 87.5 | 66.7
  Any Laboratory abnormalities: Coagulation | 25.0 | 0.0 | 33.3 | 38.9 | 10.0 | 10.0 | 35.0 | 37.8 | 36.4 | 45.5 | 37.5 | 40.0

ADVERSE EVENTS:
Time Frame: Adverse Events: Part A: First dose date up to 32 weeks plus 30 days; Part B: First dose date up to 181 weeks plus 30 days All-cause Mortality: From Study Start date (29 March 2013) up to study completion date (23 April 2019) (6 years and 1 month)
Description: The Safety Analysis Set included all participants who received at least 1 infusion at any dose level of study drug (ADX).
Arm/Group | Part A: ADX 200 mg | Part A: ADX 600 mg | Part A: ADX 1800 mg | Part B: PAC, ADX 800 mg | Part B: LAC, ADX 1200 mg | Part B: LSC, ADX 1200 mg | Part B: EGC, ADX 800 mg | Part B: FL CRC, ADX 800 mg+BEV 5 mg/kg | Part B: FL CRC, ADX 800 mg+BEV 10 mg/kg | Part B: SL CRC, ADX 800 mg+BEV 5 mg/kg | Part B: SL CRC, ADX 800 mg+BEV 10 mg/kg | Part B: BRCA, ADX 800 mg
All-Cause Mortality (participants affected / at risk) | 1/4 | 0/3 | 1/6 | 8/36 | 4/10 | 3/10 | 13/40 | 22/45 | 5/11 | 25/44 | 5/8 | 8/15
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/3 | 2/6 | 19/36 | 5/10 | 6/10 | 19/40 | 17/45 | 3/11 | 13/44 | 4/8 | 5/15
Other Adverse Events (participants affected / at risk) | 4/4 | 3/3 | 5/6 | 36/36 | 9/10 | 10/10 | 40/40 | 45/45 | 11/11 | 44/44 | 8/8 | 15/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part A: ADX 200 mg (N=4) | Part A: ADX 600 mg (N=3) | Part A: ADX 1800 mg (N=6) | Part B: PAC, ADX 800 mg (N=36) | Part B: LAC, ADX 1200 mg (N=10) | Part B: LSC, ADX 1200 mg (N=10) | Part B: EGC, ADX 800 mg (N=40) | Part B: FL CRC, ADX 800 mg+BEV 5 mg/kg (N=45) | Part B: FL CRC, ADX 800 mg+BEV 10 mg/kg (N=11) | Part B: SL CRC, ADX 800 mg+BEV 5 mg/kg (N=44) | Part B: SL CRC, ADX 800 mg+BEV 10 mg/kg (N=8) | Part B: BRCA, ADX 800 mg (N=15)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Leukocytosis (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pancytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Acute coronary syndrome (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Acute myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Atrial flutter (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Cardiac arrest (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pericardial effusion (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Adrenal haemorrhage (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Eyelid ptosis (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 2 | 0 | 0 | 0 | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Ascites (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 2 | 1 | 0 | 0 | 0 | 0
Colitis ischaemic (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 0
Duodenal obstruction (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Duodenal perforation (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Enteritis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Gastric haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Haematemesis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Ileus (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Large intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 0
Obstruction gastric (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oesophageal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Proctalgia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 3 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Catheter site extravasation (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Catheter site haematoma (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Chest pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Performance status decreased (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 5 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Hepatic failure (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Abdominal abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Bacteraemia (Infections and infestations) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Cellulitis of male external genital organ (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Cystitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Escherichia pyelonephritis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gangrene (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Influenza (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Large intestine infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Peritonitis bacterial (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 1 | 1 | 1 | 0 | 0
Pneumonia streptococcal (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pyelonephritis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rotavirus infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Sepsis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 1 | 1 | 0
Septic shock (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0
Skin infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Urosepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Carbon monoxide poisoning (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ligament sprain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Post procedural complication (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Anticoagulation drug level above therapeutic (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 3 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Failure to thrive (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Fluid overload (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Diffuse large B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Metastases to meninges (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Haemorrhage intracranial (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Transient ischaemic attack (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Tremor (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Unresponsive to stimuli (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Confusional state (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Mental status changes (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 1 | 2 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1
Haematuria (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hydronephrosis (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Urinary retention (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Urinary tract obstruction (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 2 | 1 | 1 | 0 | 0 | 0 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hypersensitivity pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 3 | 0 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1
Diabetic foot (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 2 | 0 | 0
Embolism (Vascular disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haematoma (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Shock haemorrhagic (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Part A: ADX 200 mg (N=4) | Part A: ADX 600 mg (N=3) | Part A: ADX 1800 mg (N=6) | Part B: PAC, ADX 800 mg (N=36) | Part B: LAC, ADX 1200 mg (N=10) | Part B: LSC, ADX 1200 mg (N=10) | Part B: EGC, ADX 800 mg (N=40) | Part B: FL CRC, ADX 800 mg+BEV 5 mg/kg (N=45) | Part B: FL CRC, ADX 800 mg+BEV 10 mg/kg (N=11) | Part B: SL CRC, ADX 800 mg+BEV 5 mg/kg (N=44) | Part B: SL CRC, ADX 800 mg+BEV 10 mg/kg (N=8) | Part B: BRCA, ADX 800 mg (N=15)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 11 | 7 | 2 | 12 | 9 | 1 | 11 | 2 | 3
Hypercoagulation (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Leukocytosis (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 12 | 4 | 2 | 16 | 18 | 5 | 12 | 5 | 6
Pancytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 3 | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 10 | 3 | 3 | 8 | 3 | 1 | 1 | 0 | 0
Angina pectoris (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 1
Bradycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Palpitations (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Sinus tachycardia (Cardiac disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Tachycardia (Cardiac disorders) | 0 | 0 | 0 | 3 | 1 | 0 | 1 | 2 | 0 | 0 | 0 | 0
Ear pain (Ear and labyrinth disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Tinnitus (Ear and labyrinth disorders) | 0 | 0 | 0 | 1 | 2 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 2 | 0 | 1 | 0 | 0
Conjunctival oedema (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dry eye (Eye disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 1 | 1 | 0 | 0
Erythema of eyelid (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Eye swelling (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Lacrimation increased (Eye disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 1
Ocular hyperaemia (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 1
Photopsia (Eye disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vision blurred (Eye disorders) | 0 | 0 | 0 | 2 | 1 | 0 | 2 | 1 | 0 | 1 | 0 | 1
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 2 | 0 | 1 | 2 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 0 | 1 | 4 | 4 | 0 | 2 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 1 | 6 | 0 | 2 | 5 | 12 | 1 | 11 | 5 | 3
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 4 | 5 | 1 | 3 | 1 | 1
Abdominal wall haematoma (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Anorectal discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 1 | 0
Ascites (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1
Colitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0
Constipation (Gastrointestinal disorders) | 1 | 0 | 0 | 7 | 1 | 4 | 14 | 17 | 3 | 12 | 5 | 7
Dental caries (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 2 | 0 | 0 | 16 | 4 | 2 | 19 | 25 | 3 | 28 | 6 | 5
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 6 | 4 | 1 | 1 | 0 | 1
Dyschezia (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 3 | 0 | 1 | 4 | 5 | 2 | 1 | 1 | 1
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 5 | 3 | 1 | 1 | 0 | 0
Erosive oesophagitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Flatulence (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1 | 1 | 2 | 2 | 1 | 2 | 2 | 1
Gingival bleeding (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 3 | 0 | 0
Haematochezia (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 2 | 0 | 4 | 1 | 1
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 2 | 0 | 4 | 1 | 0
Mouth ulceration (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 2 | 2 | 18 | 3 | 5 | 25 | 33 | 9 | 27 | 5 | 6
Oral pain (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 2 | 2 | 1 | 3 | 0 | 0
Proctalgia (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 6 | 1 | 0
Rectal fissure (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 4 | 0 | 2 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 2 | 0 | 7 | 11 | 1 | 15 | 4 | 1
Toothache (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0 | 2 | 9 | 1 | 2 | 13 | 14 | 5 | 14 | 3 | 2
Asthenia (General disorders) | 1 | 1 | 0 | 6 | 0 | 1 | 4 | 8 | 2 | 6 | 5 | 0
Axillary pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Catheter site pain (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Chest discomfort (General disorders) | 1 | 0 | 1 | 0 | 1 | 1 | 1 | 2 | 0 | 0 | 0 | 0
Chest pain (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 5 | 0 | 1 | 0 | 1
Chills (General disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 2 | 2 | 0 | 2 | 1 | 0
Complication associated with device (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Early satiety (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 2 | 2 | 0 | 27 | 5 | 7 | 23 | 36 | 7 | 26 | 6 | 11
Gait disturbance (General disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 3 | 4 | 1 | 1 | 0 | 0
Generalised oedema (General disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Influenza like illness (General disorders) | 0 | 0 | 0 | 3 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0
Malaise (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 0
Mucosal inflammation (General disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 5 | 8 | 0 | 9 | 0 | 1
Non-cardiac chest pain (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 3 | 1 | 1
Oedema peripheral (General disorders) | 0 | 0 | 0 | 20 | 2 | 0 | 11 | 5 | 1 | 4 | 0 | 2
Pain (General disorders) | 0 | 0 | 0 | 5 | 0 | 1 | 1 | 2 | 1 | 1 | 0 | 0
Peripheral swelling (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 2 | 1 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 8 | 1 | 1 | 6 | 2 | 0 | 8 | 2 | 0
Swelling (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Temperature intolerance (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 12 | 17 | 1 | 2 | 0 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hepatic cirrhosis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Drug hypersensitivity (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 1 | 0 | 0
Hypersensitivity (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Seasonal allergy (Immune system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0
Abscess (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bacteraemia (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Candida infection (Infections and infestations) | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 1 | 0 | 4 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 0
Cystitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Ear infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Eye infection (Infections and infestations) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastrointestinal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Hepatitis C (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Herpes zoster (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1
Hordeolum (Infections and infestations) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Infected cyst (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Laryngitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Lung infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Nail infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Nasopharyngitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 1 | 1 | 3 | 1 | 0
Oral candidiasis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 1 | 2 | 0 | 2
Pyuria (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Sinusitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 3 | 1 | 0 | 1 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 1 | 3 | 1 | 0 | 5 | 3 | 3 | 3 | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 4 | 1 | 0 | 3 | 6 | 0 | 8 | 2 | 1
Wound infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Arthropod bite (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 3 | 2 | 0 | 1 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 3 | 0 | 0 | 5 | 7 | 1 | 6 | 0 | 0
Gastrointestinal stoma complication (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 5 | 1 | 4 | 1 | 2
Injection related reaction (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Limb injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Procedural pain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Skin abrasion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Skin laceration (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 3 | 1 | 0 | 2 | 1 | 0
Stoma complication (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Wound dehiscence (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Activated partial thromboplastin time prolonged (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 4 | 1 | 4 | 0 | 3
Aspartate aminotransferase increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 1 | 2 | 6 | 1 | 3 | 1 | 3
Blood alkaline phosphatase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 1 | 1 | 0 | 1 | 1
Blood bilirubin increased (Investigations) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Blood creatinine increased (Investigations) | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 3 | 0 | 1
Blood thyroid stimulating hormone increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Carcinoembryonic antigen increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Haemoglobin decreased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Heart rate irregular (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
International normalised ratio increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 3 | 1 | 1 | 0 | 0
Liver function test increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Lymphocyte count decreased (Investigations) | 0 | 0 | 0 | 1 | 1 | 1 | 2 | 0 | 0 | 1 | 0 | 0
Neutrophil count decreased (Investigations) | 0 | 0 | 0 | 6 | 1 | 0 | 7 | 10 | 2 | 9 | 0 | 0
Platelet count decreased (Investigations) | 0 | 0 | 0 | 4 | 1 | 1 | 7 | 5 | 1 | 5 | 1 | 2
Prothrombin time prolonged (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Weight decreased (Investigations) | 0 | 0 | 0 | 7 | 0 | 0 | 5 | 7 | 1 | 1 | 1 | 0
Weight increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 2 | 0 | 0 | 1 | 0
White blood cell count decreased (Investigations) | 0 | 0 | 0 | 2 | 1 | 1 | 5 | 5 | 0 | 6 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 1 | 10 | 1 | 2 | 12 | 19 | 3 | 9 | 2 | 3
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 2 | 1 | 0 | 7 | 12 | 2 | 9 | 1 | 4
Fluid overload (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Folate deficiency (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 4 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 2 | 0 | 1 | 2 | 1 | 0 | 0 | 0 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 1 | 1 | 2 | 1 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 8 | 1 | 1 | 4 | 9 | 3 | 8 | 4 | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 3 | 0 | 0 | 1 | 3 | 0 | 5 | 2 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 3 | 0 | 1 | 3 | 2 | 0 | 0 | 0 | 1
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 2 | 1 | 0
Hypoproteinaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Malnutrition (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 2 | 0 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 1 | 0 | 3 | 6 | 10 | 1 | 8 | 0 | 3
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 2 | 1 | 1 | 7 | 9 | 1 | 3 | 2 | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 1 | 1 | 2 | 0 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 2 | 0 | 1
Joint stiffness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 2 | 1 | 3 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 3 | 0 | 1 | 4 | 3 | 0 | 4 | 0 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 2 | 1 | 0 | 1 | 2 | 0 | 1 | 0 | 2
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 4 | 8 | 1 | 4 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 7 | 0 | 3 | 2 | 3 | 0 | 5 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 8 | 0 | 1 | 5 | 4 | 0 | 4 | 2 | 1
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 3 | 0 | 1 | 0 | 0
Pathological fracture (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Spondylitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Cardiac myxoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Intracranial tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Amnesia (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Ataxia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Balance disorder (Nervous system disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Dizziness (Nervous system disorders) | 1 | 1 | 1 | 7 | 2 | 2 | 6 | 7 | 2 | 11 | 2 | 1
Dysaesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 3 | 0 | 0 | 0
Dysgeusia (Nervous system disorders) | 0 | 0 | 0 | 10 | 1 | 0 | 8 | 6 | 2 | 2 | 0 | 3
Facial paralysis (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 0 | 0 | 0 | 5 | 1 | 1 | 6 | 13 | 1 | 8 | 1 | 2
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 2 | 2 | 0 | 0 | 0 | 0
Loss of consciousness (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Memory impairment (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 1 | 0 | 0 | 0
Movement disorder (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Neuralgia (Nervous system disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Neuropathy peripheral (Nervous system disorders) | 0 | 1 | 0 | 11 | 0 | 4 | 19 | 16 | 4 | 4 | 1 | 5
Paraesthesia (Nervous system disorders) | 0 | 0 | 0 | 8 | 0 | 0 | 9 | 16 | 1 | 2 | 1 | 1
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 4 | 22 | 3 | 4 | 0 | 2
Presyncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 1 | 0
Sciatica (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Seizure (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Somnolence (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Syncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 0 | 0 | 0 | 0
Taste disorder (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 5 | 0 | 0 | 0 | 0
Toxic encephalopathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Tremor (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Vocal cord paralysis (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Agitation (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 1
Anxiety (Psychiatric disorders) | 0 | 0 | 0 | 6 | 0 | 1 | 5 | 3 | 1 | 3 | 0 | 2
Confusional state (Psychiatric disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 2 | 1 | 1 | 0 | 0
Delirium (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Depression (Psychiatric disorders) | 0 | 0 | 0 | 4 | 0 | 0 | 6 | 4 | 0 | 2 | 3 | 1
Insomnia (Psychiatric disorders) | 1 | 0 | 0 | 3 | 2 | 0 | 10 | 8 | 2 | 2 | 0 | 2
Dysuria (Renal and urinary disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 5 | 1 | 1 | 0 | 0
Haematuria (Renal and urinary disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 3 | 4 | 0 | 5 | 0 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1
Pollakiuria (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 1
Proteinuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 11 | 0 | 5 | 0 | 0
Ureterolithiasis (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Urinary incontinence (Renal and urinary disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 2 | 0 | 1 | 0 | 1
Urinary retention (Renal and urinary disorders) | 0 | 0 | 0 | 3 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 2 | 11 | 1 | 2 | 6 | 9 | 1 | 6 | 0 | 4
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 3 | 4 | 2 | 1 | 1 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 3 | 7 | 2 | 2 | 6 | 12 | 1 | 5 | 1 | 5
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 2 | 1 | 2 | 0 | 3
Emphysema (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 4 | 2 | 0 | 4 | 7 | 2 | 9 | 1 | 2
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 2 | 3 | 0 | 0 | 0 | 0 | 0 | 0
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 3 | 0 | 0 | 1 | 6 | 1 | 1 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 2 | 1 | 1 | 0 | 0
Lower respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 1 | 0 | 0 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 3 | 0 | 1 | 2 | 0 | 1 | 4 | 0 | 1
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 1
Organising pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2 | 0 | 1 | 2 | 6 | 0 | 2 | 2 | 1
Paranasal sinus hypersecretion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 0 | 0 | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 1
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 1 | 1 | 1 | 2 | 0 | 2 | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 4 | 0 | 1 | 0 | 2
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 4 | 1 | 2 | 0 | 1
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0
Sputum discoloured (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Throat tightness (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 20 | 2 | 5 | 4 | 5 | 1 | 15 | 2 | 9
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 3 | 1 | 1 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 8 | 0 | 1 | 2 | 5 | 1 | 2 | 0 | 1
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 2 | 1 | 0
Granuloma annulare (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 4 | 0 | 2 | 0 | 1
Nail discolouration (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Nail ridging (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1 | 1 | 0 | 1 | 3 | 0 | 1 | 0 | 1
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 3 | 2 | 4 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 3 | 0 | 1 | 6 | 2 | 1 | 2 | 1 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 9 | 2 | 1 | 8 | 3 | 1 | 2 | 1 | 0
Rash generalised (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rash macular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 3 | 0 | 0 | 1 | 0 | 0 | 3 | 1 | 1
Skin discolouration (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 1 | 0 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 3 | 0 | 3 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Aortic intramural haematoma (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 0 | 5 | 0 | 0 | 0 | 2 | 1 | 1 | 0 | 1
Embolism (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Flushing (Vascular disorders) | 0 | 0 | 0 | 3 | 1 | 1 | 0 | 1 | 1 | 2 | 0 | 1
Haematoma (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hot flush (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 3 | 0 | 0
Hypertension (Vascular disorders) | 1 | 0 | 0 | 3 | 0 | 0 | 2 | 18 | 2 | 5 | 0 | 0
Hypotension (Vascular disorders) | 0 | 0 | 0 | 4 | 0 | 2 | 2 | 2 | 1 | 4 | 0 | 0
Peripheral coldness (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After conclusion of the study and without prior written approval from Gilead, investigators in this study may communicate, orally present, or publish in scientific journals or other media only after the following conditions have been met:

* The results of the study in their entirety have been publicly disclosed by or with the consent of Gilead in an abstract, manuscript, or presentation form; or
* The study has been completed at all study sites for at least 2 years

DOCUMENTS (2):
  • Study Protocol (2016-08-01): https://cdn.clinicaltrials.gov/large-docs/82/NCT01803282/Prot_000.pdf
  • Statistical Analysis Plan (2019-07-24): https://cdn.clinicaltrials.gov/large-docs/82/NCT01803282/SAP_001.pdf